CLINICAL TRIAL: NCT03497234
Title: Development of a Rapid Amniotic Fluid (AF) Test and a Non-Invasive Vaginal Fluid (VF) Test to Detect Intra-Amniotic Infection and Predict Preterm Birth in Women Presenting With Preterm Labor and Intact Amniotic Membranes
Brief Title: Rapid Amniotic Fluid (AF) Test and a Non-Invasive Vaginal Fluid (VF) Test
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Strategic Decision
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D0116003
Record Dates: First submitted 2018-04-03; First posted 2018-04-13 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-04

CONDITIONS: Intra-Amniotic Infection of Foetus

STUDY DESIGN:
Intervention Model Description: This is a multi-centered, prospective study, involving pregnant women presenting to the labor and delivery unit
Masking Description: Investigator is blinded to results of the analyzer but all patients have samples run on analyzer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All women eligible to participate (Experimental): All women presenting who sign the consent and found eligible will have a VF and AF sample taken and analyzed on the Perilynx Analyzer to measure AF and VF fluid. This does not affect their regular standard of care and diagnosis
  Interventions: Diagnostic Test: Perilynx Analyzer to measure AF and VF fluid

INTERVENTIONS:
Diagnostic Test: Perilynx Analyzer to measure AF and VF fluid — Hologic developed a rapid in-vitro diagnostic system composed of an analyzer and cassettes to identify women with intra-amniotic infection.

SUMMARY:
A multi-centered, prospective study, involving pregnant women presenting to the labor and delivery unit of collaborating clinical study sites with preterm labor and intact amniotic membranes with and without suspected Intra-Amniotic Infection (IAI).

DETAILED DESCRIPTION:
A study on patients in preterm labor for whom the managing physician plans to perform amniocentesis to evaluate for possible infection using conventional, currently available methods. Vaginal fluid will be collected and analyzed and amniotic fluid will also. These tests will be run remotely and not reported to the clinician.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject has singleton gestation
3. Subject has fetus with gestational age ≥ 22 0/7 weeks and ≤ 33 6/7 weeks
4. Subject has had evidence of spontaneous preterm labor as evidenced by documented regular uterine contractions (≥4 per hour) and one or more of the following:

   1. Cervical dilation > 2cm
   2. Cervical length of ≤25 mm via transvaginal ultrasound
5. Subject has onset of contractions was within 48 hours of enrollment in the study
6. Subject has documented intact amniotic membranes
7. Subject's care provider plans to perform an amniocentesis procedure -

Exclusion Criteria:

* 1. Subject has documented ruptured amniotic membranes 2. Subject has a fetus with major fetal or genetic anomaly or chromosomal aneuploidy 3. Subject has maternal or fetal indication for preterm birth (e.g., pre-eclampsia) 4. Subject is unable to provide written informed consent 5. Subject has evidence of non-reassuring fetal heart rate tracing requiring immediate delivery 6. Subject has vaginal bleeding within the past 24 hours 7. Subject has advanced labor (cervix >4 cm dilated) 8. Subject has HIV, hepatitis 9. Subject has not been enrolled previously in this study and/or is participating in another study (that in the opinion of the Investigator) may interfere with participation in this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
performance of vaginal fluid test | 18 months
  To assess the performance of a vaginal fluid test for assessing risk of IAI in subjects presenting with preterm labor and intact membranes.
performance of amniocentesis test | 18 months
  To assess the performance of a rapid amniotic fluid test to identify intraamniotic infection (IAI).

CONTACTS AND LOCATIONS:
Overall Officials: Christina Mastandrea, Study Director — Hologic, Inc.
Locations (5):
- United States (5):
  - Good Samaritan Hospital, Long Beach, California
  - Willis Knighton, Shreveport, Louisiana
  - Rutgers, Newark, New Jersey
  - Ohio State Medical Center, Columbus, Ohio
  - Regional Obstetrical Consultants, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No